CLINICAL TRIAL: NCT06637683
Title: Multi-Strain and High-Concentration Bacillus Probiotic Spores (LiveSpo COLON) in the Supportive Treatment of Inflammatory Bowel Disease (IBD): A Blind, Randomized, and Controlled Trial
Brief Title: Efficacy of LiveSpo COLON as a Supportive Treatment for Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Vietstar Biomedical Research (Industry); Thai Binh University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COLON 01; 1015/GCN YDTB (Other: Thai Binh University of Medicine and Pharmacy)
Record Dates: First submitted 2024-09-30; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases (IBD); Bacillus spore; Crohn's disease; ulcerative colitis; adult
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: A randomized, single-blind, controlled clinical trial
Who Masked: Investigator
Masking Description: This is a single-blind study, while both patients and care providers know clearly which product is being tested, the assessor in the study is a blind assessor to ensure objectivity in the assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The Control group receives routine treatment according to the hospital's standard internal medicine protocol, which includes:
  * Anti-inflammatory drugs: sulfasalazine (Azulfidine®), corticosteroids (Prednisone)
  * Immunosuppressants: azathioprine (Imuran®) and mercaptopurine (Purinethol®)
  * Antibiotics: metronidazole (Metrogyl®)
  * Other medications: anti-diarrheal drugs, laxatives, and other pain relievers (as prescribed by a doctor).
  All concurrent medications will be documented accordingly.
  Interventions: Other: Routine treatment
- Test group (Experimental): The Experimental group receives the routine treatment and uses distilled water plus B. subtilis and B. clausii at 3 billion CFU/5 mL (LiveSpo COLON)
  The standard internal medicine treatment protocol of the hospital includes:
  * Anti-inflammatory drugs: sulfasalazine (Azulfidine®), corticosteroids (Prednisone)
  * Immunosuppressants: azathioprine (Imuran®) and mercaptopurine (Purinethol®)
  * Antibiotics: metronidazole (Metrogyl®)
  * Other medications: anti-diarrheal drugs, laxatives, and other pain relievers (as prescribed by a doctor).
  All concurrent medications will be documented accordingly.
  Interventions: Combination Product: LiveSpo COLON

INTERVENTIONS:
Combination Product: LiveSpo COLON — LiveSpo® COLON has a registration number: 10401/2019/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam
  Arms: Test group
Other: Routine treatment — The standard internal medicine treatment protocol of the hospital
  Arms: Control group

SUMMARY:
Inflammatory bowel disease (IBD) is a prevalent condition, comprising two major types: (1) Crohn disease (chronic enteritis characterized by abdominal pain, stool irregularities, fatigue, weight loss, and malnutrition) and (2) ulcerative colitis, often presenting with bloody stools. In Vietnam, approximately 20% of the population was affected by IBD, with 20% of these patients being at risk of developing colon cancer. The primary goal of treatment for IBD is to address inflammation. Various medications were found to be effective in reducing inflammation, including anti-inflammatory and antibiotic drugs. However, the use of antibiotics had a negative impact on the gut microbiota, particularly with prolonged use and increased drug resistance. In response, the supplementation of probiotics was extensively researched and applied in the prevention and treatment of ulcerative colitis and other gastrointestinal disorders over the past decade.

Oral probiotics containing Lactobacillus demonstrated lower efficacy due to reduced resilience and survival in the acidic stomach environment compared to Bacillus strains. Research suggested that supplementing with high-dose, multi-strain Bacillus probiotics could be a promising approach as supportive therapy for patients with chronic inflammatory bowel disease.

The study aimed to evaluate the effectiveness of the oral probiotic LiveSpo COLON, containing 3 billion CFU/5 mL of B. subtilis and B. clausii, as a supportive treatment for patients with chronic IBD.

Study Population: The sample size consisted of 60 patients diagnosed with ulcerative colitis at the Thai Binh University of Medicine and Pharmacy.

Study Sites: The study was conducted at the Thai Binh University of Medicine and Pharmacy, Thai Binh, Vietnam.

Description of Study Intervention: A total of 60 eligible patients were randomly divided into two groups (n = 30/group). Patients in the Control group received the conventional treatment regimen at the hospital, while those in the Experimental group (Colon group) were administered LiveSpo® Colon (3 billion CFU/5 mL) at a dose of 3 ampoules/day-one ampoule in the morning, noon, and evening-in combination with the conventional treatment regimen. All patients were monitored for 30 days, after which they continued to be observed following the protocol of the hospital.

Study Duration: 5 months.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a prevalent condition encompassing two major types: (1) Crohn disease (chronic enteritis characterized by symptoms such as abdominal pain, stool irregularities, fatigue, weight loss, and malnutrition) and (2) ulcerative colitis, often associated with bloody stools. In Vietnam, it is estimated that in 2018, about 4 million Vietnamese suffered from chronic colitis. IBD affects approximately 20% of the population, with 20% of these patients at risk of developing colon cancer. The pathogenesis of chronic IBD remains unclear. Recent studies have noted abnormalities in the gut microbiota in Crohn's disease, including an increase in pathogenic bacteria such as E. coli, Proteobacteria, and Actinobacteria, and a decrease in Firmicutes and Bacteroides.

The treatment of IBD is challenging and complex due to its progressive nature and recurring episodes. The current treatment goal for IBD is to address inflammation. Many medications help reduce inflammation, including anti-inflammatory drugs such as sulfasalazine, corticosteroids like prednisone, and immunosuppressants such as azathioprine and mercaptopurine. Metronidazole is an antibiotic that can also help eliminate bacteria in the intestines, particularly in cases of Crohn disease. Most people with chronic IBD will need to take at least one type of medication for an extended period to reduce current symptoms, prevent inflammation, and decrease the frequency of future episodes. However, some anti-inflammatory drugs or steroids can cause numerous adverse effects, such as nausea, increased risk of infections, osteoporosis, diabetes, and obesity. Additionally, the use of antibiotics can negatively impact the gut microbiota, especially with prolonged treatment and increased drug resistance. Patients with severe ulcerative colitis who do not respond to medical treatment may require surgery to remove part or all of the colon.

Probiotics are live microorganisms that can provide health benefits when consumed in adequate amounts, typically ranging from 1 to 10 billion per day, depending on the purpose of prevention or supportive treatment. The probiotic Lactobacillus plantarum L.1375 has been shown to be as effective as mesalamine, promoting the secretion of anti-inflammatory cytokines used in the treatment of Crohn's disease. However, oral probiotics containing Lactobacillus have shown lower efficacy due to their reduced resilience and survival in the acidic environment of the stomach compared to Bacillus strains. Several Bacillus species, such as B. subtilis and B. clausii, have the ability to form endospores, allowing them to withstand harsh environmental conditions like heat, acid, and bile. This means that Bacillus probiotics are more likely to survive in the harsh conditions of the gastrointestinal tract and reach the small intestines, where they can provide various health benefits. Bacillus probiotics have also demonstrated natural resistance to some antibiotics, making them a potentially more effective option for patients taking antibiotics or with a history of antibiotic use.

The objective of this study was to evaluate the safety and effectiveness of the oral probiotic LiveSpo COLON, containing 3 billion CFU/5 mL of B. subtilis and B. clausii, as a supportive treatment for patients with chronic IBD.

A randomized, blind, controlled clinical trial was conducted. Participants provided various information, including their names, ages, and antibiotic/anti-inflammatory history. After obtaining informed consent, 60 eligible patients were randomly assigned to two groups (n = 30/group) using permuted block randomization with R.3.2 software. The Control group received conventional treatment, while the Experimental group (Colon group) received LiveSpo® Colon (3 billion CFU/5 mL) at a dose of 3 ampoules/day-one ampoule in the morning, noon, and evening-in addition to the conventional treatment. All patients were monitored for 30 days, after which they continued under hospital care following standard protocol. Clinical and subclinical evaluations were performed on Days 7 and 30.

Clinical Evaluation:

- Interview: Conducted via telephone or at the research facility using the IBDQ-32 questionnaire to assess health-related quality of life in patients with IBD (ulcerative colitis and Crohn's disease). The questionnaire covered bowel symptoms (BS), systemic symptoms (SS), emotional function (EF), and social function (SF), with each question rated from 1 to 7 (1 being worst, 7 being best). Total IBDQ scores ranged from 32 to 224, assessed on Days 0, 7, and 30.

Sub-clinical Evaluation:

* Blood Tests: 13 hematological indices and 7 biochemical indices were evaluated on Day 30.
* Colonoscopy: Changes before and after treatment were assessed to evaluate lesion characteristics on colonoscopy, including redness, bleeding, swelling, and ulcers, on Days 7 and 30.

Data collection and statistical analysis involved compiling medical records and organizing patient information into a dataset. The safety and efficacy of LiveSpo COLON were evaluated by comparing the Control and Colon groups based on changes in biochemical and hematological indicators, improvement in IBD symptoms (BS, SS, EF, SF, and total scores), and improvements in colon ulcers (redness, inflammation, bleeding, swelling, and ulceration) before and after treatment.

Tabular analysis was performed on dichotomous variables using the χ² test or Fisher exact test when the expected value of any cell is below five. Continuous variables were compared using either the t-test or the Wilcoxon/Mann-Whitney test when the data were not normally distributed. Statistical and graphical analyses were conducted using SAS 9.4 software. The significance level for all analyses is set at p less than 0.05.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 years and older.
* Diagnosed with IBD based on the hospital's routine diagnostic process, which includes: (i) Positive stool test for bacteria, parasites, or fungi; (ii) Colonoscopy results showing ulcerative lesions with biopsy samples taken for histopathology; (iii) Presence of persistent gastrointestinal symptoms such as abdominal pain, stool disorders (diarrhea or constipation with mucus and blood), fatigue, and weight loss.
* Patients who have voluntarily signed the consent form to participate in the study.

Exclusion criteria:

* Patients did not have the test results and symptoms as described in the inclusion criteria; patients met the inclusion criteria but did not comply with the study procedures
* Patients who did not participate in any other clinical trial during 3 months before this study or use any probiotic product as similar as the experimental product
* Patients were indicated for surgery to treat ulcerative colitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with IBD symptoms and score representing the severity of patients' IBD symptoms in control and experiment group | Day 0 and Day 7 and Day 30
  Disease symptoms are assessed according to severity from 1-7 based on the 32-question IBDQ-32 questionnaire with 4 symptom assessment domains,including: Bowel Symptom (BS), Systemic Symptom (SS), Emotional Function (EF) and Social Function (SF). Each question is graded from 1 to 7 (1 is the worst situation and 7 is the best situation). The IBDQ total score is within the range from 32 to 224, higher score represented higher life quality.

SECONDARY OUTCOMES:
Number of patients with positive changes in colon lesions before and after treatment | Day 0 and Day 30
  Endoscopic images showing changes in colon lesions including red inflammation, bleeding, swelling and ulceration before treatment and after treatment
Number of participants with abnormal laboratory blood test results | Day 30
  Evaluate the safety of LiveSpo COLON by assessing the proportion of patients with abnormal biochemical and hematological indicators Hematological indicators: white blood cell (G/L); red blood cell (T/L); hemoglobin (g/L); Hematocrit (%); Mean corpuscular volume (fL); Mean Corpuscular Hemoglobin (pg); Mean Corpuscular Hemoglobin Concentration (g/L); Red Cell Distribution Width (%); Platelet count (G/L); Mean of hemoglobin red blood cells (pg); Red blood cell Distribution Width - Coefficient of Variation(%); Mean platelet volume (fL); Platelet volume (%).
  Biochemical indicators: Glutamate Oxaloacetat Transaminase (U/L), Glutamate Pyruvate Transaminase (U/L),Gamma-Glutamyl Transferase(G/L); Bilirubin (μmol/L): Albumin (g/L); Urea (mmol/L); Creatin (μmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen T Binh, Assoc.Prof., Principal Investigator — Thai Binh University of Medicine and Pharmacy
Locations (1):
- Thai Binh University of Medicine and Pharmacy, Thái Bình, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study report (CSR). For more information or to submit a request, please contact clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Background] Lefevre M, Racedo SM, Denayrolles M, Ripert G, Desfougeres T, Lobach AR, Simon R, Pelerin F, Justen P, Urdaci MC. Safety assessment of Bacillus subtilis CU1 for use as a probiotic in humans. Regul Toxicol Pharmacol. 2017 Feb;83:54-65. doi: 10.1016/j.yrtph.2016.11.010. Epub 2016 Nov 5. PMID 27825987
- [Background] Moayyedi P, Ford AC, Talley NJ, Cremonini F, Foxx-Orenstein AE, Brandt LJ, Quigley EM. The efficacy of probiotics in the treatment of irritable bowel syndrome: a systematic review. Gut. 2010 Mar;59(3):325-32. doi: 10.1136/gut.2008.167270. Epub 2008 Dec 17. PMID 19091823
- [Background] Lee ES, Song EJ, Nam YD, Lee SY. Probiotics in human health and disease: from nutribiotics to pharmabiotics. J Microbiol. 2018 Nov;56(11):773-782. doi: 10.1007/s12275-018-8293-y. Epub 2018 Oct 24. PMID 30353462
- [Background] Horosheva T V, Vodyanoy V, Sorokulova I. Efficacy of Bacillus probiotics in prevention of antibiotic-associated diarrhoea: a randomized double-blind, placebo-controlled clinical trial. JMM Case Reports. 2014;1(3):e004036
- [Background] Ismaeil H, Abdo W, Amer S, et al.Ameliorative Effect of Heat-Killed Lactobacillus plantarum L. 137 and/or Aloe vera against Colitis in Mice. Processes. 2020;8(2):225.
- [Background] Sadrin S, Sennoune S, Gout B, Marque S, Moreau J, Zinoune K, Grillasca JP, Pons O, Maixent JM. A 2-strain mixture of Lactobacillus acidophilus in the treatment of irritable bowel syndrome: A placebo-controlled randomized clinical trial. Dig Liver Dis. 2020 May;52(5):534-540. doi: 10.1016/j.dld.2019.12.009. Epub 2020 Jan 15. PMID 31952938
- [Background] Horosheva TV, Vodyanoy V, & Sorokulova I. Efficacy of Bacillus probiotics in prevention of antibiotic-associated diarrhoea: a randomized, double-blind, placebo-controlled clinical trial. JMM Case Reports. 2014; 1(3), e004036.
- [Background] Fisher SA, Tremelling M, Anderson CA, Gwilliam R, Bumpstead S, Prescott NJ, Nimmo ER, Massey D, Berzuini C, Johnson C, Barrett JC, Cummings FR, Drummond H, Lees CW, Onnie CM, Hanson CE, Blaszczyk K, Inouye M, Ewels P, Ravindrarajah R, Keniry A, Hunt S, Carter M, Watkins N, Ouwehand W, Lewis CM, Cardon L; Wellcome Trust Case Control Consortium; Lobo A, Forbes A, Sanderson J, Jewell DP, Mansfield JC, Deloukas P, Mathew CG, Parkes M, Satsangi J. Genetic determinants of ulcerative colitis include the ECM1 locus and five loci implicated in Crohn's disease. Nat Genet. 2008 Jun;40(6):710-2. doi: 10.1038/ng.145. Epub 2008 Apr 27. PMID 18438406
- [Background] Miele E, Pascarella F, Giannetti E, Quaglietta L, Baldassano RN, Staiano A. Effect of a probiotic preparation (VSL#3) on induction and maintenance of remission in children with ulcerative colitis. Am J Gastroenterol. 2009 Feb;104(2):437-43. doi: 10.1038/ajg.2008.118. Epub 2009 Jan 20. PMID 19174792
- [Background] Yarlas A, Maher S, Bayliss M, Lovley A, Cappelleri JC, Bushmakin AG, DiBonaventura MD. The Inflammatory Bowel Disease Questionnaire in Randomized Controlled Trials of Treatment for Ulcerative Colitis: Systematic Review and Meta-Analysis. J Patient Cent Res Rev. 2020 Apr 27;7(2):189-205. doi: 10.17294/2330-0698.1722. eCollection 2020 Spring. PMID 32377552